CLINICAL TRIAL: NCT04699487
Title: Efficacy and Safety of CareMin650 Used for the Prevention of Oral Mucositis in Patients With Head and Neck Cancer Starting Radiotherapy: the PrOMiSE Study
Brief Title: Efficacy and Safety of CareMin650 for Prevention of Oral Mucositis in HNC Patients Starting Radiotherapy
Acronym: PrOMiSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoMedLight (Industry)
Collaborators: Monitoring Force Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NML-20-01
Record Dates: First submitted 2020-12-22; First posted 2021-01-07 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer; Oral Mucositis (Ulcerative) Due to Radiation; Radiation Therapy Complication
Keywords: Photobiomodulation; Head and Neck Cancer; Oral Mucositis; Radiation Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis; Ulcer | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient receiving Photobiomodulation (Experimental)
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Oral pads will be applied on irradiated areas presenting a risk of radiotherapy-related OM. In addition, a derma pad will be applied on the anterior face of the neck to protect the oropharynx from OM.
  The dose to be delivered, at each session and each applied area, has been set at 3 J/cm². In case a lesion appears, the dose will be increased to 6J/cm² for curative treatment.
  Treatment with CareMin650 must start on the first day of radiotherapy and will be administered during the whole radiotherapy period, ideally 5 days/week, at least 3 days/week, ideally before the radiotherapy session.

SUMMARY:
Oral mucositis (OM) can affect up to 90% of head and neck cancer (HNC) patients treated with radiation therapy (RT). The Mucositis Study Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO) recommends the use of photobiomodulation (PBM) in the prevention of OM.

PBM is the application of lasers or non-coherent light sources such as LEDs, to beneficially influence cellular metabolism.

Even though PBM has proved its efficacy, this therapeutic option is currently limited by lack of standardization, accuracy and reproducibility. CareMin650 has been developed to overcome these issues, since it allows a reproducible delivery of light, independently of the operator. Additionally, it is easy to use and user-friendly.

PrOMiSE is a prospective, interventional, one-group, open-label, multicentric, international study conducted in European sites, specialized in radio-oncology.

Patients with head and neck cancer (HNC) starting RT and with no oral mucositis (OM) lesion at the time of inclusion, will be eligible. They will be treated by PBM using CareMin650 during the whole period of radiotherapy.

DETAILED DESCRIPTION:
Oral mucositis (OM) can affect up to 90% of head and neck cancer (HNC) patients treated with radiation therapy (RT) and/or chemotherapy (CT). It can be as severe as WHO grade 3 / 4 in 35% to more than 50% of cases. The pathobiology of OM relates to injuries that occur in the epithelial and connective tissues, as a response to a complex cascade of biological events, involving all the tissues and cellular elements of the mucosa (Sonis et al., 2004). OM may result in dysphagia, pain, risk of infection, weight loss, interruption or modification of anticancer therapy, or hospitalization.

As OM is a major and frequent side effect of RT, the Mucositis Study Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO) has published clinical practice guidelines for mucositis prevention secondary to cancer therapy. In addition to meticulous oral hygiene, MASCC/ISOO also suggests several therapeutic preventive strategies: growth factors, cytokines, anti-inflammatory agents, natural agents, … In the 2020 guidelines, photobiomodulation (PBM) formerly known as Low-Level Laser Therapy (LLLT), has obtain a full recommendation for the prevention of OM in patients undergoing RT, with or without concomitant CT, for HNC.

PBM is the application of lasers or non-coherent light sources such as LEDs, to beneficially influence cellular metabolism. In a Cochrane review that included 32 clinical trials, PBM was the only treatment that demonstrated a reduction in the risk of severe mucositis. In 2011, a meta-analysis included 11 placebo-controlled randomized trials in 415 patients treated with CT or RT for head and neck cancer (HNC) or hematopoietic stem cell transplantation. According to MASCC/ISOO recommendations, PBM is now recommended to prevent OM in HNC patients receiving RT with or without chemotherapy . The 2014 recommendations have been endorsed by the AFSOS (Association Française pour les Soins de Support en Oncologie) in France. Finally, the National Institute for Health and Care Excellence (NICE) determined that PBM for OM shows no major safety concerns and that evidence on efficacy is adequate in quality and quantity.

Taken together, these data show that PBM is an efficacious and safe option to prevent and/or treat radiotherapy-related OM.

Even though PBM has proved its efficacy, delivery of PBM in OM is currently limited by lack of standardization, accuracy and reproducibility. In particular, the distance between the lighting source and the mucosa or skin is difficult to assess and control accurately. Therefore, the amount of energy delivered may vary from one session to another, as well as from one operator to another.

CareMin650 has been developed to overcome these issues. CareMin650 allows a reproducible delivery of light, independently of the operator. As light is emitted by a flexible surface in contact with the mucosa or the skin, the dose delivered will be controlled. Additionally, it is meant to be easy to use and user-friendly. An interim analysis of SafePBM, a pilot study performed in France provided preliminary data on safety and efficacy. Among 186 CareMin650 sessions performed to prevent (n=152) or treat (n=34) OM in patients with HNC, no treatment-emergent adverse event was considered related to the device and no adverse event led to CareMin650 discontinuation. Only one out of 7 (14%) HNC patients treated in the preventative setting developed OM grade 3. However, this patient had started PBM 6 days after the initiation of RT, instead of starting at day 1 of RT. These encouraging results suggest that CareMin650 is both well tolerated and efficient to prevent severe OM in these high-risk patients.

The aim of the present study is to show the efficacy and safety of the CareMin650 medical device, in the prevention of severe OM in HNC patients receiving radiotherapy. The rate of severe OM will be compared to severe OM rate reported in the literature.

This is a prospective, interventional, one-group, open-label, multicentric, international study that will be conducted in Belgian and German sites, specialized in radio-oncology.

Photobiomodulation will be delivered to all included patients with the CareMin650 (NeoMedLight).

The studied Device CareMin 650 consists in a lightbox and a light applicator that delivers red light at 650nm to the oral mucosa and the neck. The applicator is composed of a connector, a fiberoptic beam of about 1 meter long and a light textile part. Appropriate non-sterile single use disposable sleeves will be added by the operator to cover the part in contact with the patient's mucosa or skin.

This device is CE marked and is used in this study in its intended indication.

No interim analysis is planned.

ELIGIBILITY:
Inclusion Criteria:

* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2.
* Histologically proven squamous cell carcinoma of oropharynx, hypo pharynx or oral cavity, with or without prior surgical resection.
* Starting intensity modulated radiation therapy (IMRT) or VoluMetric Arc Therapy (VMAT) on at least 50% of the oral mucosa at a total dose of at least 50 Gy, alone or associated with chemotherapy or targeted therapies.
* Dental examination prior to radiotherapy and any required dental treatment have been performed.

Exclusion Criteria:

* Any ongoing malignancy located in head or neck other than primary head and neck cancer (distant metastasis or extension).
* Any active cancer other than primary head and neck cancer.
* Only enteral/parenteral feeding or only liquid food intake are possible.
* Ongoing keratinocyte growth factors (palifermin) use.
* Known polyurethane allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least one OM grade >2 at any time during radiotherapy. | 5-10 weeks
  To investigate the efficacy of CareMin650 in the prevention of oral mucositis in patients with HNC starting radiotherapy.

SECONDARY OUTCOMES:
Frequency of AE classified using MedDRA dictionary | 5-10 weeks
  To investigate the safety of CareMin650
Grading of AE using CTCAE V5 | 5-10 weeks
  To investigate the safety of CareMin650
Number of patient with a temporary or sustains discontinuation of PBM due to AE | 5-10 weeks
  To investigate the safety of CareMin650
Time to OM lesions occurrence | 5-10 weeks
  To describe the patterns of OM lesions
Grade (WHO and CTCAE version 3) of OM lesions | 5-10 weeks
  To describe the patterns of OM lesions
Time to OM lesions resolution (defined as lesions that do not require further treatment) | 5-10 weeks
  To describe the patterns of OM lesions
Average duration of WHO grade 3 OM | 5-10 weeks
  To describe the duration of the grade 3 OM
Satisfaction of operators having use the device evaluated by a sponsor semi-quantitative satisfaction questionnaire. | Through study completion, an average of 1 year
  To investigate the handling and the convenience of the device from the operator's perspective
Satisfaction of the patient having use the device evaluated by a sponsor semi-quantitative satisfaction questionnaire. | Through patient study completion, an average of 2 months
  To investigate the patient satisfaction
Percentage of subject with onset of xerostomia during the study | 5-10 weeks
  To evaluate the evolution of xerostomia
Percentage of subject with onset of dysgeusia during the study | 5-10 weeks
  To evaluate the evolution of dysgeusia
Maximum severity of dysphagia as assessed by CTCAE V3 | 5-10 weeks
  To evaluate the evolution of dysphagia
Evolution of body weight over time | 5-10 weeks
  To evaluate the evolution of body weight

OTHER OUTCOMES:
For each neck dermatitis lesion: date of onset, location and CTCAE v5 grade | 5-10 weeks
  To estimate the incidence and severity of neck radiation dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Elbe, MD, Principal Investigator
Locations (1):
- UNIKLINIK RWTH AACHEN - Klinik für Radioonkologie und Strahlentherapie, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trotti A, Bellm LA, Epstein JB, Frame D, Fuchs HJ, Gwede CK, Komaroff E, Nalysnyk L, Zilberberg MD. Mucositis incidence, severity and associated outcomes in patients with head and neck cancer receiving radiotherapy with or without chemotherapy: a systematic literature review. Radiother Oncol. 2003 Mar;66(3):253-62. doi: 10.1016/s0167-8140(02)00404-8. PMID 12742264
- [Background] Elad S, Cheng KKF, Lalla RV, Yarom N, Hong C, Logan RM, Bowen J, Gibson R, Saunders DP, Zadik Y, Ariyawardana A, Correa ME, Ranna V, Bossi P; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2020 Oct 1;126(19):4423-4431. doi: 10.1002/cncr.33100. Epub 2020 Jul 28. PMID 32786044
- [Background] Antunes HS, Herchenhorn D, Small IA, Araujo CMM, Viegas CMP, de Assis Ramos G, Dias FL, Ferreira CG. Long-term survival of a randomized phase III trial of head and neck cancer patients receiving concurrent chemoradiation therapy with or without low-level laser therapy (LLLT) to prevent oral mucositis. Oral Oncol. 2017 Aug;71:11-15. doi: 10.1016/j.oraloncology.2017.05.018. Epub 2017 Jun 3. PMID 28688677
- [Background] Pulito C, Cristaudo A, Porta C, Zapperi S, Blandino G, Morrone A, Strano S. Oral mucositis: the hidden side of cancer therapy. J Exp Clin Cancer Res. 2020 Oct 7;39(1):210. doi: 10.1186/s13046-020-01715-7. PMID 33028357